CLINICAL TRIAL: NCT00659269
Title: A Randomized Phase III Study of Vitamins B6 and B12 to Prevent Chemotherapy-Induced Neuropathy in Cancer Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: INST 0553C; NCI-2012-00946 (Registry Identifier: National Cancer Institute CTRP)
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: Vitamin B-12; Vitamin B-6; Chemotherapy-Induced Neuropathy; Taxanes; Vinca alkaloid; Heavy metals; Neuropathy; Nerve pain
MeSH Terms: conditions — Neoplasms; Neuralgia | interventions — Geritol; Vitamin B 12; Vitamin B 6; Drug Therapy; Cisplatin; Oxaliplatin; Paclitaxel; Albumin-Bound Paclitaxel; Docetaxel; Vincristine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multivitamin (MV) (Active Comparator): 1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Interventions: Dietary Supplement: Multivitamin (MV); Drug: Chemotherapy
- Multivitamin + Vitamin B12 + Vitamin B6 (Experimental): 1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Interventions: Dietary Supplement: Multivitamin + Vitamin B12 + Vitamin B6; Drug: Chemotherapy

INTERVENTIONS:
Dietary Supplement: Multivitamin (MV) — Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  Arms: Multivitamin (MV)
Dietary Supplement: Multivitamin + Vitamin B12 + Vitamin B6 — Multivitamin (containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12), plus Vitamin B6 tablets and Vitamin B12 injections
  Arms: Multivitamin + Vitamin B12 + Vitamin B6
Drug: Chemotherapy — Patients are treated per standard of care according to the choice of the treating physician with heavy metals (cisplatin, oxaliplatin), taxanes (paclitaxel, docetaxel), or vinca alkaloids (vincristine, vinorelbine)
  Ranges of cumulative doses (in mg/m2) are:
  paclitaxel, 700-960; docetaxel, 240-400; vincristine, 8-16; vinorelbine, 360-480; cisplatin, 240-400; oxaliplatin, 400-800; abraxane, 1200-1800
  Other Names: Cisplatin (Platinol, Platinol-AQ); Oxaliplatin (Eloxatin); Paclitaxel (Taxol, Abraxane); Docetaxel (Taxotere); Vincristine (Oncovin); Vinorelbine tartrate (Navelbine)

SUMMARY:
Many types of chemotherapy may cause nerve damage as a side effect. This neurotoxicity can manifest as peripheral sensory neuropathy (characterized by numbness, tingling, or pain). The goal of this study is to determine the efficacy of the combination of vitamin B6 and B12 in preventing chemotherapy induced neuropathy.

DETAILED DESCRIPTION:
Neuropathy can be a significant side effect of chemotherapy using platinum compounds, taxanes, and vinca alkaloids. There is clinical and preclinical data that vitamin B6 and B12 may alleviate neuropathy in experimentally induced neuropathy in animal models, or clinical neuropathy such as diabetic neuropathy. This is a randomized phase III study of the use of multivitamins with or without vitamin B6 and B12 to prevent or relieve neuropathic toxicity from chemotherapy in patients receiving chemotherapy. Patients will be stratified by type of chemotherapy agent (3 groups), presence or absence of neuropathy at baseline, and randomized to receive placebo or vitamin B6/B12 supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18 years of age or older, with a cancer treated with any of the following drugs are eligible:

   * Taxanes, vinca alkaloid analogs, heavy metals.
   * Each patient will be allocated to the following 3 groups:

     * Group 1 (Heavy metals): Patients treated with cisplatin (>25 mg/m2/week dose intensity) or oxaliplatin
     * Group 2 (Taxane): Patients treated with paclitaxel, docetaxel or abraxane
     * Group 3 (Vinca alkaloids): Patients treated with vincristine and vinorelbine.
2. Patients must have a life expectancy of at least 24 weeks.
3. Patients must have a Zubrod performance status of 0-2.
4. Patients must sign an informed consent.
5. Patients may have a grade 0 (chemotherapy naive) or 1 neuropathy (history of prior chemotherapy) prior to entry.

Exclusion Criteria:

1. Patients with symptomatic brain metastases are excluded from this study.
2. Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
3. Patients may receive no other concurrent complementary medicines during this study.
4. Patients with neuropathy induced diabetes are not eligible for this study
5. Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2006-07; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zoneddy Dayao, MD, Principal Investigator — UNM Cancer Center
Locations (5):
- United States (5):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Cancer Center at Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico

REFERENCES:
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between July, 2006, and September, 2013, at participating cancer clinics across the state of New Mexico
Groups:
- Multivitamin (MV): Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
- Multivitamin + Vitamin B12 + Vitamin B6: Multivitamin, plus Vitamin B6 tablets and Vitamin B12 injections
  Multivitamin + Vitamin B12 + Vitamin B6: As in Arm 1, one multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Cumulative doses (in mg/m2) are:
  paclitaxel, 700; docetaxel, 300; vincristine, 16; navelbine, 480; cisplatin, 300; oxaliplatin, 400
Period: Overall Study
Arm/Group | Multivitamin (MV) | Multivitamin + Vitamin B12 + Vitamin B6
Started | 157 | 162
Group 1 (Heavy Metals) | 52 | 52
Group 2 (Vinca Alkaloids) | 12 | 12
Group 3 (Taxanes) | 92 | 97
Completed | 156 | 161
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multivitamin (MV) | Multivitamin + Vitamin B12 + Vitamin B6 | Total
Number analyzed (Participants) | 157 | 162 | 319
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 83] | 54.5 [18 to 80] | 55 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 116 | 230
  Male | 43 | 46 | 89
Region of Enrollment [Number; unit: participants]
  United States | 157 | 162 | 319

OUTCOME MEASURES:

1. Primary Outcome: Neurotoxicity Assessment at Baseline
Description: Neurotoxicity is evaluated using The Functional Assessment of Cancer Therapy-Taxane (FACT-Tax) questionnaire. FACT-Tax is a validated, self-reported instrument. The questionnaire consists of 11 questions and possible scores for each question range from 0 (no neurotoxicity symptoms) to 4 (worst possible neurotoxicity symptoms). The total score for any patient can therefore range from 0 to 44. The questionnaire is given to patients to fill out at baseline (prior to chemotherapy treatment) and the mean total score for all patients is reported.
Time Frame: At study start; prior to treatment (week 0)
Population: Of the 92 and 97 patients in the MV arm and MV + Vit.B12 + VitB6 arm, 84 and 86 patients, respectively, in the Group 1 (Taxanes) completed the FACT-Tax questionnaire at baseline and the analysis is presented here. This also applies to 48 and 45 patients in Group 2 (Heavy Metals) and 10 and 12 patients in Group 3 (Vincas)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Taxane Group: Multivitamin (MV) Arm: Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Ranges of cumulative doses (in mg/m2) are:
  paclitaxel, 700-960; docetaxel, 240-400; abraxane, 1200-1800
- Taxane Group: MV + Vitamin B12 + Vitamin B6: Multivitamin (MV) plus Vitamin B6 tablets and Vitamin B12 injections
  Multivitamin + Vitamin B12 + Vitamin B6: As in Arm 1, one multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Ranges of cumulative doses (in mg/m2) are:
  paclitaxel, 700-960; docetaxel, 240-400
- Heavy Metals Group: Multivitamin (MV) Arm: Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Cumulative doses for chemotherapy (in mg/m2) are:
  cisplatin, 240-400; oxaliplatin, 400-800
- Heavy Metals Group: MV + Vitamin B12 + Vitamin B6 Arm: Multivitamin (MV) plus Vitamin B6 tablets and Vitamin B12 injections
  Multivitamin + Vitamin B12 + Vitamin B6: As in Arm 1, one multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Ranges of cumulative doses (in mg/m2) are:
  cisplatin, 240-400; oxaliplatin, 400-800
- Vinca Alkaloids Group: Multivitamin (MV) Arm: Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Cumulative doses for chemotherapy (in mg/m2) are:
  vincristine, 8-16; vinorelbine, 360-480
- Vinca Alkaloids Group: MV + Vitamin B12 + Vitamin B6 Arm: Multivitamin (MV) plus Vitamin B6 tablets and Vitamin B12 injections
  Multivitamin + Vitamin B12 + Vitamin B6: As in Arm 1, one multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Ranges of cumulative doses (in mg/m2) are:
  vincristine, 8-16; vinorelbine, 360-480
Arm/Group | Taxane Group: Multivitamin (MV) Arm | Taxane Group: MV + Vitamin B12 + Vitamin B6 | Heavy Metals Group: Multivitamin (MV) Arm | Heavy Metals Group: MV + Vitamin B12 + Vitamin B6 Arm | Vinca Alkaloids Group: Multivitamin (MV) Arm | Vinca Alkaloids Group: MV + Vitamin B12 + Vitamin B6 Arm
Number analyzed (Participants) | 84 | 86 | 48 | 45 | 10 | 12
units on a scale | 8.5 (8.5) | 7.3 (7.3) | 5.23 (5.86) | 4.58 (5.34) | 6.80 (5.09) | 2.08 (2.02)

2. Primary Outcome: Neurotoxicity Assessment at Cycle 2
Description: Neurotoxicity is evaluated using The Functional Assessment of Cancer Therapy-Taxane (FACT-Tax) questionnaire. FACT-Tax is a validated, self-reported instrument. The questionnaire consists of 11 questions and possible scores for each question range from 0 (no neurotoxicity symptoms) to 4 (worst possible neurotoxicity symptoms). The total score for any patient can therefore range from 0 to 44. The questionnaire is given to patients to complete at completion of cycle 2 of chemotherapy treatment and the mean total score for all patients is reported.
Time Frame: 2 weeks
Population: Of the 92 & 97 patients in the MV and MV + Vit.B12 + VitB6 arms, 72 & 80 patients, respectively, in the Group 1 (Taxanes) both completed 2 cycles of treatment and completed the FACT-Tax questionnaire at cycle 2, and the analysis is presented here. The same applies to 27 & 25 patients in Group 2 (Heavy Metals) and 9 & 10 patients in Group 3 (Vinca)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Taxane Group: MV + Vitamin B12 + Vitamin B6: Multivitamin, plus Vitamin B6 tablets and Vitamin B12 injections
  Multivitamin + Vitamin B12 + Vitamin B6: As in Arm 1, one multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Ranges of cumulative doses (in mg/m2) are:
  paclitaxel, 700-960; docetaxel, 240-400; abraxane, 1200-1800
- Heavy Metals Group: Multivitamin (MV) Arm: Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Ranges of cumulative doses (in mg/m2) are:
  cisplatin, 240-400; oxaliplatin, 400-800
- Vinca Alkaloids Group: Multivitamin (MV) Arm: Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Ranges of cumulative doses (in mg/m2) are:
  vincristine, 8-16; vinorelbine, 360-480
Arm/Group | Taxane Group: Multivitamin (MV) Arm | Taxane Group: MV + Vitamin B12 + Vitamin B6 | Heavy Metals Group: Multivitamin (MV) Arm | Heavy Metals Group: MV + Vitamin B12 + Vitamin B6 Arm | Vinca Alkaloids Group: Multivitamin (MV) Arm | Vinca Alkaloids Group: MV + Vitamin B12 + Vitamin B6 Arm
Number analyzed (Participants) | 72 | 80 | 27 | 25 | 9 | 10
units on a scale | 13.0 (10.9) | 12.0 (9.9) | 9.7 (5.99) | 8.4 (7.16) | 14.56 (12.9) | 5.6 (6.59)

3. Primary Outcome: Neurotoxicity Assessment at Cycle 4
Description: Neurotoxicity is evaluated using The Functional Assessment of Cancer Therapy-Taxane (FACT-Tax) questionnaire. FACT-Tax is a validated, self-reported instrument. The questionnaire consists of 16 questions and possible scores for each question range from 0 (no neurotoxicity symptoms) to 4 (worst possible neurotoxicity symptoms). The total score for any patient can therefore range from 0 to 44. The questionnaire is given to patients to fill out at completion of cycle 4 of their chemotherapy treatment and the mean total score for all patients is reported.
Time Frame: 4 weeks
Population: Of the 92 & 97 patients in the MV and MV + Vit.B12 + VitB6 arms, 57 & 65 patients, respectively, in Group 1 (Taxanes) completed both 4 cycles of chemotherapy and completed the FACT-Tax questionnaire at cycle 4, and the analysis is presented here. The same applies to 28 & 21 patients in Group 2 (Heavy Metals) and 6 & 9 patients in Group 3 (Vinca)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Multivitamin + Vitamin B12 + Vitamin B6: Multivitamin (MV) plus Vitamin B6 tablets and Vitamin B12 injections
  Multivitamin + Vitamin B12 + Vitamin B6: As in Arm 1, one multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts).
  The patient will also take the following, starting on the first day of chemotherapy:
  1. pyridoxine 50 mg three times per day, orally and continue for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  2. Vitamin B12 one mg injected intramuscularly, every 3 or 4 weeks, depending on the timing of the chemotherapy for 4 doses.
  Ranges of cumulative doses (in mg/m2) are:
  paclitaxel, 700-960; docetaxel, 240-400; abraxane, 1200-1800
Arm/Group | Taxane Group: Multivitamin (MV) Arm | Multivitamin + Vitamin B12 + Vitamin B6 | Heavy Metals Group: Multivitamin (MV) Arm | Heavy Metals Group: MV + Vitamin B12 + Vitamin B6 Arm | Vinca Alkaloids Group: Multivitamin (MV) Arm | Vinca Alkaloids Group: MV + Vitamin B12 + Vitamin B6 Arm
Number analyzed (Participants) | 67 | 58 | 28 | 21 | 6 | 9
units on a scale | 14.5 (11.4) | 14.5 (11.1) | 8.71 (6.5) | 7.05 (6.55) | 17.5 (5.36) | 9.22 (10.22)

4. Primary Outcome: Change in Neurotoxicity Assessment Between Cycle 4 and Baseline
Description: Neurotoxicity is evaluated using The Functional Assessment of Cancer Therapy-Taxane (FACT-Tax) questionnaire. FACT-Tax is a validated, self-reported instrument. The questionnaire consists of 11 questions and possible scores for each question range from 0 (no neurotoxicity symptoms) to 4 (worst possible neurotoxicity symptoms). The total score for any patient can therefore range from 0 to 44. The questionnaire is given to patients to fill out at baseline, cycle 2, and cycle 4 of their chemotherapy treatment. Change in neurotoxicity scores from baseline to the completion of 4 cycles are reported as the mean total score for all patients.
Time Frame: 4 weeks
Population: Of the 92 & 97 patients in the Multivitamin (MV) and MV + Vit.B12 + VitB6 arms, 54 & 62, respectively, in Group 1 (Taxanes) completed both 4 cycles of chemo and the FACT-Tax questionnaire at baseline and cycle 4; analysis is presented here. The same applies to 28 & 20 patients in Group 2 (Heavy Metals) and 5 & 9 patients in Group 3 (Vinca)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Taxane Group: Multivitamin (MV) Arm: Multivitamin only
  Multivitamin (MV): Multivitamins containing no more than 10 mg of pyridoxine and/or 10 micrograms of Vitamin B12 will be given to the patients on this arm.
  1 multivitamin pill will be taken orally, daily starting on the first day of chemotherapy and continuing for no more than 30 days past the cumulative chemotherapy dose (until the next cycle starts)
  Ranges of cumulative doses (in mg/m2) are:
  paclitaxel, 700-960; docetaxel, abraxane, 1200-1800
Arm/Group | Taxane Group: Multivitamin (MV) Arm | Taxane Group: MV + Vitamin B12 + Vitamin B6 | Heavy Metals Group: Multivitamin (MV) Arm | Heavy Metals Group: MV + Vitamin B12 + Vitamin B6 Arm | Vinca Alkaloids Group: Multivitamin (MV) Arm | Vinca Alkaloids Group: MV + Vitamin B12 + Vitamin B6 Arm
Number analyzed (Participants) | 54 | 62 | 28 | 20 | 5 | 9
units on a scale | 7.0 (9.9) | 7.2 (9.8) | 3.9 (7.1) | 4.7 (5.7) | 11.8 (4.7) | 7 (9.2)
Statistical Analysis 1: Comparison: Taxane Group: Multivitamin (MV) Arm vs Taxane Group: MV + Vitamin B12 + Vitamin B6; Test type: Superiority or Other; p = 0.91, ANOVA

ADVERSE EVENTS:
Description: Since vitamin B6 and B12 are food supplements with only rare toxic effects, no toxicity will be recorded. Only serious adverse (SAE) will be reported, whether or not related to these vitamins.
Arm/Group | Multivitamin (MV) | Multivitamin + Vitamin B12 + Vitamin B6
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/162
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The number of completed surveys decreased as time went on for each group of patients. This resulted in small numbers of patients to analyze, especially in Group 3 (Vinca Alkaloids), since there weren't many patients in this group to begin with.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes